CLINICAL TRIAL: NCT01790321
Title: Efficacy Study of Water as Fortification Vehicle for Zinc for Improving Zinc Status in Primary Schools Children in the Municipality of Natitingou, North of Benin.
Brief Title: Water-based Zinc Efficacy Trial in Beninese Shool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Michael B. Zimmermann (Other)
Collaborators: Université d'Abomey-Calavi (Other)
Responsible Party: Sponsor-Investigator, Prof. Michael B. Zimmermann, Prof. Dr.med, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LSF_Zn_school
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Zinc Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pump water (No Intervention): Untreated pump water (pump water recognised as improved water source by WHO)
- Filtered water (Placebo Comparator): Pump water purified by the LSF-filtering device
  Interventions: Device: LSF-filtering device
- Zinc water (Experimental): Pump water purified and zinc-fortified by the LSF-filtering device
  Interventions: Device: LSF-filtering device

INTERVENTIONS:
Device: LSF-filtering device — LifeStraw Family is a water purification device that by means of hollow fibres removes solid particles (<0.5 NTU turbidity reduction), bacteria (>Log 6 reduction), viruses (>Log 4 reduction) and cysts (>Log 3 reduction). Zinc fortification is provided by a chamber housing a zinc releasing glass-plate that is placed annexed to the hollow fibre column. It is estimated that the LSF can provide about 5 mg of zinc/l of filtered water. By consuming daily a portion of 0.6 litres of enriched water, >100% of the age-specific estimated physiologic requirement would be covered, assuming a fractional absorption of 40%.
  Other Names: LifeStraw Family by Vestergaard Frandsen SA
  Arms: Filtered water; Zinc water

SUMMARY:
The general objective of this study is to determine the effect of the daily consumption of zinc-fortified water provided by the LSF-filter on zinc status and diarrhea rates in school age children from rural areas characterized by a high risk of zinc deficiency and by elevated stunting prevalence.

DETAILED DESCRIPTION:
A double-blind efficacy study will be carried out over 4 months in school age children enrolled in a primary school equipped with a water pump, in the rural area of the commune of Natitingou, Benin. Participating children will be randomly assigned to one of two groups of intervention or control. On a daily basis, all children will consume a defined quantity of pump-water outside of meals. The water offered to children in the first group of intervention will be previously filtered and zinc-fortified by the LSF-filter; the children in the second group will receive water that has been filtered only. A nutrition survey will provide an indication of dietary zinc intake. The effect of enriched water consumption on children's zinc status will be evaluated by analyzing the concentration of zinc in serum at baseline, midpoint and endpoint of the intervention. Diarrhea rates will be monitored by recording episodes of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* School aged children enrolled in primary school and regularly attending class

Exclusion Criteria:

* Severe anemia (Hb < 7 g/dl)
* Consumption of a supplement or dietary supplement containing zinc
* Use of drugs that affect the metabolism of zinc
* Suffering from a chronic disease affecting the metabolism of zinc

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Zinc status | Baseline, midpont (varying between weeks 5-20), endpoint (week 22)
  Serum zinc concentration

SECONDARY OUTCOMES:
Inflammation status | Baseline, midpoint (varying between weeks 5-20), endpoint (week 22)
  Concentration of CRP in serum
Iron status | Baseline, midpoint (varying between weeks 5-20), endpoint (week 22)
  Haemoglobin level
Diarrhea incidence | Weekly, from baseline through to endpoint
  Occurrence of diarrhea episodes monitored over 2 days weekly
Malaria prevalence | Baseline, midpoint (varying between weeks 5-20), endpoint (week 22)
  Screening of HRP-II antigen
ALRI prevalence | At baseline and endpoint
  Auscultation and respiratory frequence (no. of chest movements per minute)
Anthropometric indices | Baseline, midpoint (varying between weeks 5-20), endpoint (week 22)
  Measurement of height, weight and mid-upper arm circumference for the assessment of height-for-age, weight-for-age and BMI-for-age Z-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr.med, Study Chair — ETH Zurich
Locations (1):
- Kotopounga primary school, Natitingou, Atakora Department, Benin

REFERENCES:
- [Derived] Galetti V, Mitchikpe CE, Kujinga P, Tossou F, Hounhouigan DJ, Zimmermann MB, Moretti D. Rural Beninese Children Are at Risk of Zinc Deficiency According to Stunting Prevalence and Plasma Zinc Concentration but Not Dietary Zinc Intakes. J Nutr. 2016 Jan;146(1):114-23. doi: 10.3945/jn.115.216606. Epub 2015 Nov 25. PMID 26609168
- [Derived] Galetti V, Kujinga P, Mitchikpe CE, Zeder C, Tay F, Tossou F, Hounhouigan JD, Zimmermann MB, Moretti D. Efficacy of highly bioavailable zinc from fortified water: a randomized controlled trial in rural Beninese children. Am J Clin Nutr. 2015 Nov;102(5):1238-48. doi: 10.3945/ajcn.115.117028. Epub 2015 Oct 14. PMID 26468121